CLINICAL TRIAL: NCT01356550
Title: A Study on The Effect of Hepatic Impairment on The Pharmacokinetics of RO4917838
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BP25260; 2010-023641-30 (EudraCT Number)
Record Dates: First submitted 2011-05-18; First posted 2011-05-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (2):
- Healthy subjects (Experimental)
  Interventions: Drug: RO4917838
- Hepatic impairment (Experimental)
  Interventions: Drug: RO4917838

INTERVENTIONS:
Drug: RO4917838 — single oral dose

SUMMARY:
This open-label, single-dose, parallel group study will assess the pharmacokinetics and safety of RO4917838 in healthy volunteers and patients with mild, moderate or severe chronic hepatic impairment. Patients and healthy volunteers will receive a single oral dose of RO4917838.

ELIGIBILITY:
Inclusion Criteria:

General:

* Body mass index (BMI) between 18 and 32 kg/m2 inclusive

Healthy Subjects:

* Adult male or female subjects, 18-70 years of age

Hepatically impaired patients:

* Adult patients, 18-65 years of age
* Documented chronic stable mild/moderate/severe liver disease (Child-Pugh class A, B or C)
* Hepatic impairment should be primary and must not be a complication of an underlying primary disease

Exclusion Criteria:

General:

* Pregnant or lactating women
* Suspicion of drug abuse or addiction at time of screening/Day -1 or history of drug abuse in the last month (patients) or last year (healthy volunteers) prior to Day -1
* Confirmed significant allergic reactions against any drug, or multiple allergies in the judgement of the investigator
* Positive for HIV infection
* Renal insufficiency

Healthy volunteers:

* History of significant disease, or evidence of disease or condition which could interfere with the study or relapse during or immediately after the study
* Any history of depressive episodes or treatment with antidepressants
* Alcohol consumption averaging more than 2 units (16 g) of alcohol for females or 3 units (24 g) for males per day, or positive alcohol breath test at screening/Day -1
* Positive for hepatitis B and/or hepatitis C infection

Hepatically impaired patients:

* Evidence of unstable clinically significant disease other than impaired hepatic function, or condition or disease which could interfere with the study or relapse during or immediately after the study
* Episode of acute depression within the last 6 months or current or previous (within the last 6 months) antidepressant treatment
* Hepatocellular carcinoma or acute hepatic disease caused by infection or drug toxicity
* Presence of surgically created or transjugular intrahepatic portal systemic shunts
* Biliary liver cirrhosis or other causes of hepatic impairment not related to parenchyma disorder and/or disease of the liver

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of RO4917838 (area under the concentration-time curve, Cmax) | 22 days

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Rennes, France
- Moscow, Russia